CLINICAL TRIAL: NCT04239313
Title: Phase Ib Clinical Trial Evaluating the Safety and Immunogenicity of Freeze-dried Recombinant Tuberculosis Vaccine (AEC / BC02) in Healthy Adults
Brief Title: A Phase Ib Study of the Recombinant Mycobacterium Tuberculosis Vaccine Freeze-dried (AEC/BC02)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AEC/BC02-Ⅰb-healthy
Record Dates: First submitted 2020-01-16; First posted 2020-01-27 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Vaccine
MeSH Terms: conditions — Tuberculosis | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Population I (Experimental): Population I has 10 subjects,and it is considered as Tuberculin purified protein derivative(TB-PPD) skin test and specific gamma-interferon (γ-IFN) detection result all negative.Population I are coxal muscle injection of low dose vaccine.
  Interventions: Biological: Low-dose freeze-dried recombinant tuberculosis vaccine (AEC / BC02)
- Population II (Active Comparator): Population I has 10 subjects,and it is considered as Tuberculin purified protein derivative(TB-PPD) skin test and specific gamma-interferon (γ-IFN) detection result all negative.Population I are coxal muscle injection of low dose adjuvant.
  Interventions: Biological: Low-dose adjuvant for freeze-dried recombinant tuberculosis vaccine (AEC / BC02)
- Population III (Placebo Comparator): Population I has 10 subjects,and it is considered as Tuberculin purified protein derivative(TB-PPD) skin test and specific gamma-interferon (γ-IFN) detection result all negative.Population I are coxal muscle injection of placebo.
  Interventions: Biological: Lyophilized recombinant tuberculosis vaccine (AEC / BC02) placebo

INTERVENTIONS:
Biological: Low-dose freeze-dried recombinant tuberculosis vaccine (AEC / BC02) — Population I are coxal muscle injection of low dose vaccine.
  Arms: Population I
Biological: Low-dose adjuvant for freeze-dried recombinant tuberculosis vaccine (AEC / BC02) — Population I are coxal muscle injection of low dose adjuvant.
  Arms: Population II
Biological: Lyophilized recombinant tuberculosis vaccine (AEC / BC02) placebo — The placebo drug contains 20mg mannitol and 10 millimole(mM) phosphate buffer(PB).population I are coxal muscle injection of placebo.
  Arms: Population III

SUMMARY:
Single-center, single-dose, placebo-controlled, open-label trials were used to evaluate the safety and immunogenicity of low-dose adjuvants and low-dose vaccines in the upper arm deltoid muscle intramuscularly in the double negative population. Thirty (PPD-QFT-) healthy adult subjects aged 18-45 were selected and divided into placebo group, low-dose adjuvant group, and low-dose vaccine group. During the test, each subject must not change groups and inoculate drugs. Every two weeks (0-2-4-6-8-10 weeks), alternately inject a dose of placebo or left and right upper arm deltoid muscles. Low-dose adjuvant or low-dose vaccine, a total of 6 doses.

DETAILED DESCRIPTION:
Single-center, single-dose, placebo-controlled, open-label trials were used to evaluate the safety and immunogenicity of low-dose adjuvants and low-dose vaccines in the upper arm deltoid muscle intramuscularly in the double negative population. Thirty (PPD-QFT-) healthy adult subjects aged 18-45 were selected and divided into placebo group, low-dose adjuvant group, and low-dose vaccine group. During the test, each subject must not change groups and inoculate drugs. Every two weeks (0-2-4-6-8-10 weeks), alternately inject a dose of placebo or left and right upper arm deltoid muscles. Low-dose adjuvant or low-dose vaccine, a total of 6 doses.

Collected adverse events within 14 days after each dose of vaccination, non-recruited adverse events within 30 days after the first dose of vaccination, subjects will receive 6 months follow-up after the last dose of vaccination, and study throughout Serious adverse events were recorded during the period. Immunogenicity will be assessed before the first dose, 24 hours after the third dose, before the fourth dose, 24 hours after the sixth dose, 1 month, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age 18-45 years old, body mass index (BMI) = weight (kg) / [(height (m) × (height (m))], in the range of 18.0 to 29.9 (including the boundary value);
* (2) I agree to participate in this study and sign an informed consent, and I am willing and able to comply with the requirements of the clinical research protocol;
* (3) Vital signs (reference range of vital signs: systolic blood pressure 90 ~ 140mmHg (including boundary value), diastolic blood pressure 60 ~ 90mmHg (including boundary value), pulse rate 50 ~ 100 beats / min (including boundary value), body temperature (ear Temperature) 35.4 ~ 37.7 ℃ (including the boundary value)), physical examination, clinical laboratory (blood routine, urine routine, blood biochemistry, hepatitis B and AIDS syphilis examination, etc.), electrocardiogram and abdominal B-ultrasound examination, the results showed no abnormalities or abnormalities Non-clinical significance
* (4) Chest X-ray examination showed no abnormalities;
* (5) TB-PPD skin test induration average diameter <5mm and QFT negative test results;
* (6) No contraindications to vaccination and no history of TB exposure.

Exclusion Criteria:

* (1) (Ask) Suffering from acute disease, severe chronic disease, acute episode of chronic disease, acute infectious disease, such as: treatment of malignant tumor, autoimmune disease, progressive atherosclerosis or diabetes with complications, Chronic obstructive pulmonary disease, acute or progressive liver or kidney disease, congestive heart failure, etc. that require oxygen therapy;
* (2) (Ask) those with eczema or other skin diseases;
* (3) (Ask) Those who are known to be allergic to the components of the test drug;
* (4) (Ask) those who have a clear diagnosis of tuberculosis, extrapulmonary tuberculosis or tuberculosis has been cured;
* (5) (Ask) a history of convulsions, epilepsy, encephalopathy and neurological symptoms or signs;
* (6) (Ask) long-term use of antibiotics;
* (7) (Ask) People with known or suspected immune function impairment or abnormality, such as those who received immunosuppressant or immune enhancer treatment within 3 months, received gastrointestinal within 3 months Those who have immunoglobulin preparations or blood products or plasma extracts outside the tract, those with human immunodeficiency virus infection or related diseases;
* (8) (inquiry) those who have no spleen, functional spleen, and spleen or splenectomy caused by any situation
* (9) Examination of one or more clinical significance of hepatitis B surface antigen, hepatitis C virus antibody, anti-human immunodeficiency virus antibody or anti- Treponema pallidum specific antibody;
* (10) Those who have a history of drug abuse or are positive for drug screening;
* (11) Those who donated or lost blood more than 400mL within 3 months before screening;
* (12) those with acute febrile diseases and infectious diseases;
* (13) those who are pregnant, lactating, or have a positive pregnancy test before vaccination, or who cannot guarantee contraception during the study period of this clinical trial;
* (14) Participated in other new drug clinical trials 3 months before screening;
* (15) Any situation that the investigator believes may affect the eva

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
The number of adverse events after intramuscular injection | Up to 6 months after the sixth time injection
  The adverse events observed mainly from laboratory examination(including vital signs/routine blood/routingurine/Liver and kidney fuction/Electrocardiograghy and Chest X-ray detection),skin reactivity and local reaction after drug injection.Vital signs(breathing,pulse,blood pressure,body temperature) of each volunteer before each dose injection,and 30min after injection.Routine blood,routine urine,liver and kidney function,and ECG before first dose,fourth dose,and 7 days after the sixth time injection;skin reactivity and local reaction of rach volunteer at 30min before and after every injection.

SECONDARY OUTCOMES:
Laboratory markers of immunity | Up to 6 months after the sixth time injection
  Evaluation of IFN-γand antibody level of before and after the immune,intracellular cytokine staining in blood .

CONTACTS AND LOCATIONS:
Overall Officials: Zhaolin Huang, Principal Investigator — Wuhan infectious disease hospital
Locations (1):
- Wuhan Infectious Disease Hospital, Wuhan, Hubei, China

REFERENCES:
- [Background] Pulendran B, Ahmed R. Immunological mechanisms of vaccination. Nat Immunol. 2011 Jun;12(6):509-17. doi: 10.1038/ni.2039. PMID 21739679
- [Background] Mostowy S, Onipede A, Gagneux S, Niemann S, Kremer K, Desmond EP, Kato-Maeda M, Behr M. Genomic analysis distinguishes Mycobacterium africanum. J Clin Microbiol. 2004 Aug;42(8):3594-9. doi: 10.1128/JCM.42.8.3594-3599.2004. PMID 15297503
- [Derived] Li J, Fu L, Guo X, Yang Y, Dong J, Wang G, Zhao A. Novel BC02 Compound Adjuvant Enhances Adaptive and Innate Immunity Induced by Recombinant Glycoprotein E of Varicella-Zoster Virus. Vaccines (Basel). 2022 Dec 15;10(12):2155. doi: 10.3390/vaccines10122155. PMID 36560565